CLINICAL TRIAL: NCT07337785
Title: Clinical Study on the Safety, Efficacy, and Pharmacokinetics of Universal CAR-T Cell Injection Targeting CD19/BCMA in Patients With Neurological Autoimmune Diseases
Brief Title: CD19/BCMA-Targeted UCAR-T for Patients With Neurological Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daishi Tian (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Daishi Tian, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD06-05-NI-01
Record Dates: First submitted 2025-12-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Relapsing or Refractory Multiple Sclerosis (MS); Myasthenia Gravis (MG); Chronic Inflammatory Demyelinating Polyneuropathy (CIDP); Autoimmune Encephalitis (AE)
MeSH Terms: conditions — Recurrence; Multiple Sclerosis; Myasthenia Gravis; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Intervention Model Description: This is a single-group assignment design. All eligible participants undergo lymphodepleting chemotherapy followed by a single intravenous infusion of RD06-05. The trial includes multiple disease cohorts (MS, MG, AE, and CIDP), but all participants receive the same intervention without randomization or comparator arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART Treatment Group (Experimental): Participants receive lymphodepleting chemotherapy with fludarabine and cyclophosphamide from Day -5 to Day -3, followed by a single intravenous infusion of RD06-05.
  Interventions: Biological: CD19/BCMA-targeted CAR-T cells; Drug: Lymphodepleting Conditioning

INTERVENTIONS:
Biological: CD19/BCMA-targeted CAR-T cells — Participants will receive lymphodepleting chemotherapy with fludarabine and cyclophosphamide followed by a single intravenous infusion of CD19/BCMA-targeted CAR-T cells (RD06-05) at dose of 1 × 10^7 CAR+ T cells/kg (Additional dose levels will be determined by safety, PK/PD, and preliminary efficacy).
  Other Names: RD06-05
Drug: Lymphodepleting Conditioning — From Day -5 to Day -3 prior to cell infusion (Day 0), subjects will receive chemotherapy preconditioning based on the "Fludarabine + Cyclophosphamide" (FC regimen). The recommended preconditioning regimen is as follows:
  Fludarabine: 30 mg/m² per day, once daily for 3 consecutive days; Cyclophosphamide: 300 mg/m² per day, once daily for 3 consecutive days;

SUMMARY:
This single-arm, open-label investigator-initiated trial (IIT) evaluates the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of RD06-05 in patients with autoimmune neurological diseases, including Multiple Sclerosis (MS), Myasthenia Gravis (MG), Chronic Inflammatory Demyelinating Polyneuropathy (CIDP), Autoimmune Encephalitis (AE), and other B-cell-mediated neuroautoimmune disorders.

In this study, the dose of CAR-T cells administered is 10×10⁶ CAR⁺T cells per kilogram of body weight. Investigators may decide whether to add other dose groups based on the subjects' safety data, pharmacokinetic (PK) data, pharmacodynamic (PD) data, and preliminary efficacy data.

For each indication, 6 to 9 subjects will be enrolled, with a total of 24 to 36 subjects planned for enrollment in the entire study.

ELIGIBILITY:
General Inclusion Criteria for All Participants:

1. Patients voluntarily agree to participate in this trial and sign the informed consent form.
2. Aged ≥ 18 years and ≤ 70 years, regardless of gender.
3. Organ function and laboratory test requirements:

   1. Liver function: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3 × Upper Limit of Normal (ULN); Total Bilirubin (TBIL) ≤ 2 × ULN (except for patients with Gilbert's syndrome).
   2. Renal function: Serum creatinine ≤ 1.5 × ULN OR creatinine clearance rate ≥ 40 ml/min.
   3. Complete blood count: Neutrophil count ≥ 1 × 10⁹/L; hemoglobin ≥ 60 g/L; platelet count ≥ 20 × 10⁹/L; lymphocyte count > 0.3 × 10⁹/L.
   4. Coagulation function: International Normalized Ratio (INR) ≤ 1.5 × ULN OR Prothrombin Time (PT) ≤ 1.5 × ULN.
   5. Oxygen saturation (SpO₂) ≥ 92% at rest while breathing room air.
   6. Echocardiography shows Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
4. For female patients of childbearing potential at screening, the result of serum or urine pregnancy test is negative.
5. Female of childbearing potential must use effective contraception from at least 28 days before apheresis until 12 months after RD06-05 infusion. Male of reproductive potential must use effective barrier contraception during the same period and must not donate semen or sperm throughout the study.

Specific Inclusion Criteria for Patients with MS:

1. Diagnosed as Relapsing-Remitting Multiple Sclerosis (RRMS), Primary Progressive Multiple Sclerosis (PPMS), or Secondary Progressive Multiple Sclerosis (SPMS) by a neurologist with diagnostic and treatment qualifications in accordance with the 2017 Revised McDonald Criteria, and relevant diagnostic documents must be provided.
2. Expanded Disability Status Scale (EDSS) score ranging from 3.0 to 7.5 (inclusive of the cutoff values).
3. Having undergone a brain MRI examination that meets the 2017 McDonald Criteria within 12 months prior to screening (must include T2/FLAIR and gadolinium-enhanced T1 sequences), showing spatial multiplicity (≥ 2 typical MS lesion regions) and/or temporal multiplicity (new T2 or gadolinium-enhanced [Gd+] lesions).
4. Previous cerebrospinal fluid (CSF) examination or CSF examination report during the screening period indicating at least one of the following conditions:

   1. Elevated IgG index
   2. Detection of one or more IgG oligoclonal bands (OCB)
5. Having received high-efficacy disease-modifying therapy (DMT) for at least 6 months, with the occurrence of any of the following conditions during the treatment period:

   1. Clinically confirmed relapse by a neurologist (new or recurrent persistent neurological deficit lasting ≥ 24 hours, excluding other causes such as fever/infection)
   2. EDSS progression (defined as: an increase of ≥ 1.0 point if EDSS ≤ 5.5; or an increase of ≥ 0.5 point if EDSS > 5.5) High-efficacy DMTs include but are not limited to: anti-CD20 monoclonal antibodies (e.g., Ocrelizumab), lymphocyte-depleting therapies (e.g., Alemtuzumab, Cladribine), and α4 integrin blockers (e.g., Natalizumab).
6. RRMS patients must meet one of the following criteria: at least 1 documented relapse within 1 year prior to screening, or at least 2 documented relapses within 2 years prior to screening, or brain MRI indicating active gadolinium-enhanced lesions or new T2 lesions within 1 year prior to screening. PPMS or SPMS patients must have documented evidence of disability progression within 2 years prior to screening. All relapses or MRI activity must be supported by medical records (e.g., outpatient/inpatient records, MRI reports, EDSS assessment forms).

Specific Inclusion Criteria for Patients with MG:

1. Meet the diagnostic criteria for generalized myasthenia gravis (gMG) in line with international myasthenia gravis (MG) consensus guidelines (e.g., the 2020 Myasthenia Gravis Foundation of America [MGFA] Guidelines).
2. Classified as MGFA Clinical Class II, III, or IV (per the MGFA Clinical Classification system for myasthenia gravis).
3. Serological testing at screening shows positivity for acetylcholine receptor antibodies (AChR-Ab), muscle-specific tyrosine kinase antibodies (MuSK-Ab), or low-density lipoprotein receptor-related protein 4 antibodies (LRP4-Ab); or there is a documented history of positivity for AChR-Ab, MuSK-Ab, or LRP4-Ab in previous medical records.
4. Score of ≥ 6 points on the Myasthenia Gravis Activities of Daily Living (MG-ADL) Scale, with the score related to ocular symptoms accounting for less than 50% of the total score.
5. Score of ≥ 8 points on the Quantitative Myasthenia Gravis (QMG) Score, with ≥ 4 items each scoring at least 2 points.
6. Having received at least one of the following treatments prior to screening, with relevant medical documentation provided:

   1. Immunosuppressants (including but not limited to azathioprine, mycophenolate mofetil, methotrexate, cyclosporine, tacrolimus, cyclophosphamide, etc.)
   2. Biologic agents (including but not limited to complement C5 inhibitors, FcRn blockers, etc.).
7. As judged by the investigator, the subject has received stable current treatment for MG for at least 3 months and has experienced any of the following:

   1. An increase of ≥ 2 points in the total MG-ADL score, with an increase of ≥ 1 point in non-ocular items;
   2. An increase of ≥ 3 points in the total QMG score, or an increase of ≥ 1 point in each of ≥ 2 non-ocular muscle items;
   3. Need for increased medication dosage, hospitalization, or emergency intervention due to MG exacerbation.

Definition of "stable treatment":

i). If the subject is taking acetylcholinesterase inhibitors, they must have received treatment with a stable dosage and regimen for at least 2 weeks prior to screening; ii). If the subject is using glucocorticoids, they must have received treatment with a stable dosage and regimen for at least 2 weeks prior to screening; iii). If the subject is receiving biologics, complement inhibitors, or FcRn blockers, they must have received treatment with a stable dosage for at least 4 weeks prior to screening; iv). If the subject is receiving other immunosuppressants or small-molecule targeted therapeutic agents, they must have received treatment with a stable dosage for at least 2 weeks prior to screening; v). If glucocorticoids and/or immunosuppressants were discontinued prior to screening due to intolerance or lack of efficacy, the discontinuation must have occurred at least 4 weeks before screening.

Specific Inclusion Criteria for Patients with CIDP:

1. Diagnosed as progressive or relapsing chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) or meeting the criteria for possible CIDP in accordance with the 2021 Guidelines of the European Academy of Neurology (EAN)/Peripheral Nerve Society (PNS), with supporting evidence including at least the following: electrophysiological findings (slowed nerve conduction velocity in ≥ 2 nerves + conduction block/temporal dispersion), elevated cerebrospinal fluid (CSF) protein level (> 45 mg/dL), nerve root thickening on MRI, or nerve biopsy results (if applicable).
2. CIDP Disease Activity Status (CDAS) score ≥ 2 at screening.
3. Inflammatory Neuropathy Cause and Treatment (INCAT) score ≥ 2 at screening: For patients with an INCAT score of 2, the score must be entirely from lower limb function; for patients with an INCAT score ≥ 3, there is no requirement on whether the score comes from upper or lower limbs.
4. Having received any of the following treatments for at least 3 months, with either the INCAT score improves by < 2 points compared to the baseline, or the treatment discontinuation due to adverse reactions:

   1. Intravenous immunoglobulin (IVIG): ≥ 2 g/kg per course, with at least 2 courses completed;
   2. Oral prednisone: ≥ 0.5 mg/kg per day for 3 months;
   3. Plasma exchange: ≥ 5 sessions per course, with at least 1 course completed;
   4. FcRn blockers (e.g., Efgartigimod): ≥ 1 full treatment cycle completed.
5. If receiving glucocorticoid treatment, the subject must have received stable dosage and regimen for at least 2 weeks before screening; if receiving immunosuppressants or small-molecule targeted therapeutic drugs, the subject must have received stable dosage for at least 2 weeks before screening.

Inclusion Criteria for AE Patients:

1. According to the 2016 International Diagnostic Criteria for Autoimmune Encephalitis (AE), the patient is clinically diagnosed with autoimmune encephalitis and meets all the following requirements: Positive result in the detection of at least one relevant autoantibody; Poor symptom control or intolerance to previous standardized treatment with glucocorticoids and at least one immunosuppressant/immunomodulator (including CD20 monoclonal antibody); Occurrence of an autoimmune encephalitis attack within 3 months before signing the informed consent form; At the time of screening, the disability status meets either a modified Rankin Scale (mRS) score of ≥ 2 or a Clinical Assessment Scale in Autoimmune Encephalitis (CASE) score of ≥ 4.

Exclusion Criteria:

1. Primary diagnosis of an autoimmune disease different from the study disease, which the investigator believes may confound the efficacy evaluation of the study disease.
2. Comorbidity with other clinically significant central nervous system (CNS) diseases or pathological changes prior to screening, including but not limited to: cerebrovascular accident, aneurysm, epilepsy, convulsions/seizures, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
3. History of allogeneic bone marrow or stem cell transplantation, or solid organ transplantation (e.g., kidney, lung, heart, liver), or planned future transplantation of such organs/cells.
4. For MG patients: Uncontrolled myasthenic crisis within 2 weeks prior to screening.
5. For CIDP patients: Pure sensory CIDP.
6. Presence of clinically significant cardiovascular dysfunction within 12 months prior to screening, including but not limited to: New York Heart Association (NYHA) Class III or IV heart failure, myocardial infarction, unstable angina pectoris, uncontrolled or symptomatic atrial arrhythmia, or any ventricular arrhythmia.
7. Presence of significant pulmonary or cardiac manifestations (e.g., pericarditis, pleural effusion) at screening, which the investigator assesses as making the patient unsuitable for participation in this study.
8. Patients with severe asthma or chronic obstructive pulmonary disease (COPD); patients with mild or moderate asthma or COPD receiving stable treatment are eligible for enrollment.
9. History of malignancy within 5 years prior to signing the ICF, except for fully treated or surgically resected non-melanoma skin cancer or carcinoma in situ (e.g., cervical cancer, bladder cancer, breast cancer) with no residual disease.
10. Pregnant or lactating females.
11. History of recurrent infections requiring hospitalization and intravenous antibiotics (e.g., 3 or more infections of the same type within the past year).
12. Active infection requiring systemic treatment (e.g., infectious pneumonia, tuberculosis) within 2 weeks prior to lymphodepletion.
13. Positive for hepatitis B surface antigen (HBsAg); or positive for hepatitis B core antibody (HBcAb) with positive hepatitis B virus (HBV) DNA detection in peripheral blood; positive for hepatitis C virus (HCV) antibody with positive HCV RNA in peripheral blood; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis antibody.
14. Vaccination with live-attenuated vaccines within 4 weeks prior to lymphodepletion, or planned vaccination with live-attenuated vaccines during the study.
15. Receipt of high-dose corticosteroids (prednisone ≥ 60 mg/day or equivalent dose) within 4 weeks prior to lymphodepletion, or inability to taper prednisone to ≤ 20 mg/day gradually within 3 days prior to lymphodepletion.
16. Inability to taper or discontinue background treatment gradually prior to lymphodepletion chemotherapy, as described in Table 3.
17. Receipt of plasma exchange, immunoadsorption, or intravenous immunoglobulin (IVIG) treatment within 4 weeks prior to screening.
18. A history of allergy or intolerance to calcineurin inhibitors used previously.
19. Receipt of renal replacement therapy within 3 months prior to screening, or expected need for renal replacement therapy during the study.
20. History of drug or alcohol abuse within 1 year prior to screening.
21. History or evidence of suicidal ideation within 6 months prior to screening, or any suicidal behavior within the previous 12 months, with the investigator determining a significant suicide risk.
22. Use of other investigational drugs within 4 weeks or 5 half-lives (whichever is longer) prior to screening.
23. A history of hypersensitivity or life-threatening reactions to any component or formulation of the study drug or study treatment (including lymphodepletion chemotherapy). For detailed information on the components of the study drug, please refer to the Investigator's Brochure (IB).
24. Any other condition deemed by the investigator to potentially affect study participation, pose a safety risk to the patient, or potentially confound the interpretation of study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
The incidence rates of Treatment-Emergent Adverse Events (TEAEs) | From the start of cell infusion to 24 months after infusion
Serious Adverse Events (SAEs) | From the start of cell infusion to 24 months after infusion
The incidence rate of Adverse Events of Special Interest (AESI) | From the start of cell infusion to 24 months after infusion

SECONDARY OUTCOMES:
MS:Time to first relapse; Annual Relapse Rate (ARR) | Day 14, Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 18, and Month 24 post infusion
MS: The number of new or enlarged T2 lesions on MRI during the study; | Day 14, Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 18, and Month 24 post infusion
MS: The number of newly emerged gadolinium-enhancing lesions on MRI | Day 14, Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 18, and Month 24 post infusion
MS: The change in Expanded Disability Status Scale (EDSS) score from baseline during the study | Day 14, Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 18, and Month 24 post infusion
MG: Changes in Myasthenia Gravis Activities of Daily Living Scale (MG-ADL) scores compared to baseline | At Week 12, and Months 6, 12, 18, and 24 post infusion
MG: Changes in Quantitative Myasthenia Gravis Score (QMG) scores compared to baseline | At Week 12, and Months 6, 12,18, and 24 post infusion
MG: The proportion of patients with a change of ≥2 points in MG-ADL scores | Months 12 and 24 post infusion
MG: The proportion of patients with a change of ≥3 points in Myasthenia Gravis Composite Scale (MGC) score | Months 12 and 24 post infusion
MG: Changes in the titer of MG serum-specific autoantibodies compared to baseline | Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 18, and Month 24 post infusion
CIDP: Changes in Inflammatory Neuropathy Cause and Treatment disability scale (INCAT) score compared to baseline | At Week 12, and Months 6, 12, 18, and 24 post infusion
CIDP: Changes in Inflammatory Rasch-Built Overall Disability Scale (I-RODS) score compared to baseline | Day 14, Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 18, and Month 24 post infusion
CIDP: Changes in average grip strength compared to baseline | Day 14, Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 18, and Month 24 post infusion
CIDP: Changes in Medical Research Council Scale (MRC) score compared to baseline | Day 14, Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 18, and Month 24 post infusion
Changes from baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | Months 6, 12, 18, and 24 post infusion
Changes from baseline in the Health Assessment Questionnaire - Disability Index (HAQ-DI) | Months 6, 12, 18, and 24 post infusion
Peak expansion (Cmax) | Days 0, 4, 7, 10, Day 14, Day 28, Week 8, Week 12, Month 6, Month 9, Month 12, Month 18, and Month 24 post infusion
Area under the curve (AUC₀-₂₈) | Days 0, 4, 7, 10, 14, 21, and Day 28 post infusion.
AE: Changes in CASE score from baseline | Months 6, 12, 18, and 24 post infusion
AE: Changes in MoCA scores from baseline | Month 6, 12, 18, and 24 post infusion
Changes in CGI score from baseline | Month 6, 12, 18, and 24 post infusion
AE: Changes in GCS score from baseline | Month 6, 12, 18, and 24 post infusion
Changes in MMSE score from baseline | Monthe 6, 12,18, and 24 post infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No